CLINICAL TRIAL: NCT05159271
Title: Efficacy and Safety of Azeol Nasal Spray Versus Placebo in the Treatment of Early Symptoms of Common Cold in Adults: the EXSPRAY Trial
Brief Title: Efficacy and Safety of Azeol Nasal Spray Versus Placebo in the Treatment of Early Symptoms of Common Cold in Adults
Acronym: EXSPRAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larena SAS (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEC19217
Record Dates: First submitted 2021-11-16; First posted 2021-12-16 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azeol spray nasal group (Experimental): Azéol Spray Nasal is a nasal spray. The constituents responsible for achieving the intended action are: Bifidobacterium breve LA 708, extract of cypres Cupressus sempervirens L., extract of Leguminosae Glycyrrhiza glabra L., glycerin and mannitol.
  Interventions: Device: Azeol spray nasal
- Placebo group (Placebo Comparator): The control product is a placebo with the same characteristics of appearance and packaging as Azéol Spray Nasal without the active ingredients
  Interventions: Device: Placebo nasal spray

INTERVENTIONS:
Device: Azeol spray nasal — Azeol Spray Nasal is a nasal spray intended to reduce the nasal congestion due to rhinitis, rhinosinusitis and colds which is marketed. The ID is conforming to the European Union (EU) legislation and is bearing the CE-mark. The ID is manufactured by PILEJE S.A.S (France).
  Arms: Azeol spray nasal group
Device: Placebo nasal spray — with the same characteristics of appearance and packaging as Azéol Spray Nasal without the active ingredients
  Arms: Placebo group

SUMMARY:
The main objective is to evaluate the efficacy of Azéol Spray Nasal, taken two times a day, versus placebo on nasal congestion in subject with common cold.

DETAILED DESCRIPTION:
This study is designed as a multicentric, randomized, double-blind, placebo-controlled with two-arm parallel groups clinical trial. 144 subjects presenting with early symptoms of common cold will be recruited for this study, according to the defined inclusion and exclusion criteria. The main objective is to evaluate the efficacy of Azéol Spray Nasal (Bifidobacterium breve LA 708, extract of cypres Cupressus sempervirens L., extract of Leguminosae Glycyrrhiza glabra L., glycerin and mannitol), taken two times a day, versus placebo on nasal congestion in subject with common cold.

ELIGIBILITY:
Inclusion Criteria:

I1. Subject aged between 18 and 65 years (limits included); I2. Subjects with early symptoms of common cold (onset less than or equal to 48 hours before inclusion upon subjects' declaration);

I3. Subjects with:

* A minimum nasal congestion score (blocked nose) of 2 (moderate) according to a 4-point scale (0 not present; 1 mild; 2 moderate; and 3 severe) assessed by Likert scale,
* Presenting a minimum of two common cold symptoms (runny nose, blocked nose, sore throat, and/or cough) at inclusion visit (V1) assessed with a score ≥ 1 according to a 4-point scale (0 not present; 1 mild; 2 moderate; and 3 severe) assessed by Likert,
* Minimum plugged nose (nasal congestion) score of 3 (≥ 3) assessed by WURSS-21;

I4. For women:

* Non menopausal with the same reliable contraception since at least 2 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicide gel, any oral contraceptive, intrauterine device, subcutaneous contraceptive implant, vaginal ring, surgical intervention (bilateral tubal ligation or ovariectomy or hysterectomy), ESSURE system),
* Menopausal without or with hormone replacement therapy; I5. Subject with good general and mental health according to the investigator opinion: no clinically significant and relevant abnormalities of medical history or physical examination; I6. Subject able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form; I7. Subject affiliated with a social security scheme; I8. Subject who agree to be registered on the volunteers in biomedical research file.

Exclusion Criteria:

E1. Subjects with nasal polyps/polyposis or nasal septum malformations or other nasal structural abnormalities that would compromise administration of the nasal spray (based on the declaration of the subjects); E2. Subjects with any other acute ear, nose, and throat and respiratory tract disease than the common cold (eg, tonsillitis, otitis, bronchitis) and chronic sinusitis or allergic rhinitis; E3. Subject suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, or other chronic respiratory trouble, etc.);

E4. Subject under:

* Concomitant treatment that might impair the trial results (eg, decongestants, local anesthetics, topical corticosteroids, saline solution) during the seven days prior to enrollment in the trial,
* Cough treatment or NSAID or any other treatment for the common cold during the seven days prior to enrollment in the trial,
* Any dietary supplement or probiotic; E5. Subjects with known or suspected hypersensitivity to the investigational device ingredients or to ingredients which could cause crossed allergia as cypress, peach or citrus fruit; E6. Subjects not fully vaccinated against SARS-CoV-2 virus; E7. Subjects positive for SARS-CoV-2 tested by rapid antigen test at V1; E8. Subjects with fever ≥ 38 °C; E9. Pregnant or lactating women or intending to become pregnant within the month ahead and during the whole study;

E10. Having a lifestyle deemed incompatible with the study according to the investigator as described below:

* Consuming more than 2 standard drinks of alcoholic daily or 14 weekly or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Smoking more than five cigarettes daily or more than 60 mg of nicotine daily,
* Practicing high level of physical activity (defined as more than 10 hours of intense physical activity a week, walking excluded); E11. Subject taking part in another clinical trial or being in the exclusion period of a previous clinical trial; E12. Subject having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros; E13. Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision; E14. Subject presenting a psychological or linguistic inability to sign the informed consent;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
relief of nasal congestion at 2 days | 2 days
  change from baseline in the relief of nasal congestion defined by "plugged nose", after 2 days of product intake, assessed at end of day after both spraying sessions with the "plugged nose" question

SECONDARY OUTCOMES:
relief of nasal congestion | 7 days
  Change from baseline in the relief of nasal congestion, assessed at the end of each day after both spraying sessions with a patient questionnaire
Area Under the Curve for sick feeling score, global severity score, symptom score and for quality-of-life score | 7 days
  Area Under the Curve for sick feeling score, global severity score, symptom score and for quality-of-life score, assessed at the end of each day after both spraying sessions with a patient questionnaire
Area Under the Curve for common cold symptoms | 7 days
  Area Under the Curve for common cold symptoms assessed at the end of each day after both spraying sessions with a patient questionnaire
Area Under the Curve for nine quality-of-life items | 7 days
  Area Under the Curve for nine quality-of-life items (Think clearly; Sleep well; Breathe easily; Walk, climb stairs, exercise; Accomplish daily activities; Work outside the home; Work inside the home; Interact with others; Live your personal life), assessed at the end of each day after both spraying sessions with a patient questionnaire
Area Under the Curve for the total nasal airway resistance to airflow | First day
  Area Under the Curve for the total nasal airway resistance to airflow using the rhinomanometry after treatment at day 1
Time to onset of subjective relief nasal congestion from day 1 | 7 days
  relief of symptoms defined when symptom absent is declared for plugged nose with a patient questionnaire
Time to onset of subjective relief symptoms from day 1 | 7 days
  relief of symptoms defined when symptom absent is declared for all symptoms with a patient questionnaire
Subject's assessment of common cold feeling compared to the day before | 7 days
  item 21 of a patient questionnaire (WURSS-21)
Subjects' assessment of efficacy | 7 days
  evaluated at the end of trial visit with a patient's satisfaction questionnaire
Presence of secondary infections in the month after the D7 | 1 month after D7
  assessed by investigator

OTHER OUTCOMES:
Presence of cold viruses in nasal fluid samples | 3 days
  Viral load (change from baseline) on Day 3 for various virus types and number of subjects with cleared viral infections
Safety endpoint | First day and 3 days
  The hemodynamic parameters, resting Heart Rate, Systolic Blood Pressure and Diastolic Blood Pressure
Safety endpoint | 1 month after D7
  Frequency of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CEN Nutriment, Dijon
  - Biofortis - Unité d'investigation clinique, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No
IPD won't be shared